CLINICAL TRIAL: NCT07043218
Title: A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of Universal CAR-T Cell in Patients With CD19 and/or CD20 Positive Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia.
Brief Title: A Clinical Study Exploring Universal CAR-T Cell in Patients With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Aibin Liang，MD，Ph.D., Principal Investigator, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT119X-CG11004
Record Dates: First submitted 2025-06-22; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: CT119X
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells（ chimeric antigen receptor T cells） (Experimental): CT1190B-P and CT1192 cells infusion
  Interventions: Drug: Chimeric Antigen Receptor T Cells (CAR-T)

INTERVENTIONS:
Drug: Chimeric Antigen Receptor T Cells (CAR-T) — chimeric antigen receptor T cells

SUMMARY:
A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT119X(including CT1190-P and CT1192) CAR-T Cell therapy, in Patients with Relapsed/Refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose exploratory clinical study to evaluate the safety, efficacy, cellular pharmacokinetics, and pharmacodynamics of CT119X (including CT1190-P and CT1192)cells in patients with B-ALL. It is planned to enroll 6-36participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily sign the informed consent form (ICF) and must be willing and be able to adhere to the study visit schedule and other protocol requirements
2. 18-75 years old;
3. Histologically or cytologically confirmed B-ALL;
4. Previously received at least 2 lines of systemic therapy;
5. Expected survival > 12 weeks;
6. Eastern Cooperative Oncology Group (ECOG) score 0-2;
7. Female participants of childbearing potential must have a negative pregnancy test at screening and prior to receiving preconditioning therapy。Both male and Female are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment and are absolutely prohibited from donating sperm donation or eggs for 1 year after receiving study treatment infusion during the study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Has HIV, syphilis infection, active hepatitis B virus infection (HBsAg positive and HBV-DNA above the detection limit), or active hepatitis Cvirus infection (HCV antibody and HCV-DNA positive);
3. Has any current uncontrolled active infection, including but not limited to participants with active tuberculosis (investigator 's judgment);
4. Participants' toxicities caused by previous treatment did not recover to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade1, except alopecia and other events that are judged tolerable by the investigator;
5. Patients with isolated extramedullary lesions;
6. Vaccination with live attenuated vaccines, inactivate vaccines or RNA vaccines within 4 weeks prior to informed consent;
7. Participants who are allergic or intolerant to preconditioning drugs, tocilizumab, or have other previous history of severe allergy such as anaphylactic shock;
8. Patients with heart disease in the 6 months prior to screening;
9. Presence of a second primary malignancy requiring treatment or not in complete remission within the past 2 years;
10. Serious pulmonary diseases that are judged by the investigator to potentially endanger the patient's life when participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
MTD and/or dose range | Up to 28 days after CAR-T cells infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT119X infusion
Adverse Events (AE) after CT119X infusion | 12 months after CT119X infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria

SECONDARY OUTCOMES:
Overall response rate （ORR） | Evaluate at 4, 8, 12 weeks and 6,9,12month after CAR-T infusion
  The proportion of patients with complete remission（CR）/partial response (PR) after CT119X infusion.
Complete response rate (CRR) | 12 months after CT119X infusion
  The proportion of patients with complete response(CR) after CT119X infusion
Duration of remission(DOR) | 12 months after CT119X infusion
  Participants achieving CR/PR will be included in the analysis set for DOR. DOR is defined as the time from the date of confirmed response until the date of disease relapse or death from any cause, whichever occurs first.
Time to response (TTR) | 12 months after CT119X infusion
  The time from cell infusion to the first assessment of CR or PR
Time to complete response (TTCR) | 12 months after CT119X infusion
  The time from cell infusion to the first assessment of CR
Progression-free survival (PFS) | 12 months after CT119X infusion
  The time from the infusion of CT119X cells to the first assessment of disease progression or death.
Overall survival (OS) | 12 months after CT119X infusion
  defined as the time from the date of receiving the infusion to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang MD,Ph.D., Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No